CLINICAL TRIAL: NCT06642337
Title: Effectiveness of Nutritional Educational Program on Caregiver's Knowledge and Performance Versus Oral Iron Therapy Alone on Hemoglobin Level Among Children With Iron Deficiency Anemia
Brief Title: Nutritional Educational Program On Therapy in Iron Deficiency Anemia
Acronym: NEPOT-IDA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, AMANJ YASSIN HAMAD AMIN, MSc In Pediatric Nursing, Hawler Medical University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: HawlerMUErbil
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Iron Deficiency Anemia (IDA); Nutrition Disorders; Growth Retardation
Keywords: Iron Deficiency Anemia; Pediatric Anemia; Oral Iron Therapy; Nutritional Education; Caregiver Knowledge; Hemoglobin Levels
MeSH Terms: conditions — Anemia, Iron-Deficiency; Nutrition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Education (Experimental): Participants in this arm will receive a Nutritional Educational Program designed specifically for caregivers of children diagnosed with iron deficiency anemia. This program includes a series of interactive sessions that focus on the following key components:
  Understanding Iron Deficiency Anemia: Caregivers will learn about the causes, symptoms, and health implications of iron deficiency anemia in children.
  Nutritional Education: The program will provide comprehensive information on identifying and incorporating iron-rich foods into the child's diet, including meats, leafy greens, legumes, and fortified cereals.
  Enhancing Iron Absorption: Caregivers will be educated on dietary strategies to improve iron absorption, such as consuming vitamin C-rich foods alongside iron sources and avoiding inhibitors like calcium and certain beverages during meals.
  Meal Planning and Preparation: Practical guidance will be given on how to effectively plan and prepare meals that are rich in iron and other
  Interventions: Other: Educational program +Oral Iron therapy
- Oral Iron Therapy (Experimental): Participants in this arm will receive oral iron therapy as the standard treatment for iron deficiency anemia. The intervention will include the following components:
  Prescription of Oral Iron Supplement: Participants will be prescribed a specific oral iron formulation, such as ferrous sulfate, ferrous fumarate, or ferrous gluconate, according to established clinical guidelines tailored to the child's age and severity of anemia.
  Dosage and Administration: Caregivers will receive clear instructions regarding the appropriate dosage, which will be determined based on the child's weight and medical needs. Administration guidelines will include taking the iron supplement on an empty stomach for optimal absorption, unless otherwise advised by a healthcare provider.
  Monitoring of Adherence and Response: Caregivers will be instructed on the importance of adherence to the prescribed regimen, with scheduled follow-up visits to monitor hemoglobin levels and assess the child's overall health and r
  Interventions: Other: Educational program +Oral Iron therapy

INTERVENTIONS:
Other: Educational program +Oral Iron therapy — The Nutritional Education Program is a structured intervention designed to enhance caregivers' understanding of nutrition and improve dietary practices for children suffering from iron deficiency anemia. The program comprises six weekly workshops lasting 1.5 hours each, focusing on essential topics such as the importance of iron in child development, identifying and preparing iron-rich foods, and practical meal planning strategies. Participants will engage in hands-on cooking demonstrations and receive educational materials, including recipe cards and meal planning tools, to support their learning. Knowledge assessments will be conducted at the beginning and end of the program to measure improvements in caregivers' nutritional knowledge.
  Other Names: Nutritional Education Program

SUMMARY:
The goal of this clinical trial is to evaluate whether a Nutritional Educational Program for caregivers can improve their knowledge and performance in managing iron deficiency anemia (IDA) in children, compared to oral iron therapy alone. The study focuses on children with IDA, particularly in [age range 1-5 years], and aims to determine if combining nutritional education with oral iron therapy has a greater impact on improving hemoglobin levels than iron therapy alone.

The main questions it aims to answer are:

1. Does caregiver education improve children's hemoglobin levels more effectively than oral iron therapy alone?
2. Does nutritional education improve caregiver knowledge and practices regarding iron-rich diets? Researchers will compare children who receive both caregiver education and oral iron therapy to those receiving only oral iron therapy to assess differences in hemoglobin levels.

Participants will:

Receive oral iron supplements. Caregivers will participate in educational sessions on dietary strategies to manage IDA.

DETAILED DESCRIPTION:
This clinical trial aims to explore the effectiveness of a Nutritional Educational Program for caregivers, in combination with oral iron therapy, on improving hemoglobin levels in children with iron deficiency anemia (IDA). Iron deficiency is a leading cause of anemia in children, and oral iron supplementation is the standard treatment. However, dietary habits and caregiver knowledge also play a significant role in managing this condition. This study will evaluate whether equipping caregivers with nutritional education enhances the outcomes of oral iron therapy.

The study will involve two groups of children with confirmed iron deficiency anemia:

Intervention Group: Children receiving oral iron therapy combined with a structured Nutritional Educational Program for their caregivers. The educational program will cover:

Understanding iron deficiency anemia and its effects on child health. Identification of iron-rich foods and dietary strategies to enhance iron absorption (e.g., vitamin C-rich foods).

Avoidance of dietary inhibitors that reduce iron absorption (e.g., calcium-rich foods and tea during meals).

Guidance on meal preparation and frequency to optimize iron intake. Control Group: Children receiving only oral iron therapy without the nutritional education component.

The primary outcome will be the change in hemoglobin levels over a specified period. Secondary outcomes will include caregivers' knowledge and performance, measured through pre- and post-intervention questionnaires, as well as adherence to the treatment regimen and dietary recommendations.

Participants will attend follow-up visits where hemoglobin levels will be monitored, and caregivers will be assessed for their understanding and application of the nutritional guidance provided. Data on the children's dietary intake will also be collected and analyzed.

This trial aims to determine if caregiver-focused nutritional education improves the management of IDA more effectively than iron therapy alone, potentially leading to better long-term health outcomes in children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1 year to 5 years.
2. Confirmed diagnosis of iron deficiency anemia (hemoglobin <11 g/dL).
3. A responsible caregiver must provide written informed consent for participation.
4. No acute or chronic illnesses affecting study outcomes.
5. Reside in the study area with access to participating healthcare facilities.

Exclusion Criteria:

1. Any child who has received iron supplementation or blood transfusions in the past 3 months.
2. Diagnosis of any anemia other than iron deficiency anemia.
3. Known severe allergic reactions to iron supplements.
4. Caregivers unable or unwilling to comply with study protocols.
5. Current use of medications affecting iron metabolism.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin Levels | 3 months (Measured at baseline and at the conclusion of the study).
  His outcome measure aims to assess the difference in hemoglobin levels in children diagnosed with iron deficiency anemia at the beginning of the study compared to their levels at the end of the intervention. The study will compare the effectiveness of oral iron therapy alone versus oral iron therapy combined with a Nutritional Educational Program provided to caregivers. Hemoglobin levels will be evaluated through blood tests, providing a quantitative assessment of the interventions' impact on anemia.

SECONDARY OUTCOMES:
Improvement in Caregivers' Knowledge of Iron-Rich Foods | Before the educational intervention and 3 months post-intervention.
  This measure will evaluate the change in caregivers' knowledge regarding dietary management of iron deficiency anemia before and after the Nutritional Educational Program. The assessment will be conducted using a validated questionnaire that gauges understanding of iron-rich foods, dietary sources, and practices that enhance iron absorption.

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University/College of nursing, Erbil, Kurdistan Region, Iraq, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandra J, Dewan P, Kumar P, Mahajan A, Singh P, Dhingra B, Radhakrishnan N, Sharma R, Manglani M, Rawat AK, Gupta P, Gomber S, Bhat S, Gaikwad P, Elizabeth KE, Bansal D, Dubey AP, Shah N, Kini P, Trehan A, Datta K, Basavraja GV, Saxena V, Kumar RR. Diagnosis, Treatment and Prevention of Nutritional Anemia in Children: Recommendations of the Joint Committee of Pediatric Hematology-Oncology Chapter and Pediatric and Adolescent Nutrition Society of the Indian Academy of Pediatrics. Indian Pediatr. 2022 Oct 15;59(10):782-801. PMID 36263494
- [Background] da Silva Lopes K, Yamaji N, Rahman MO, Suto M, Takemoto Y, Garcia-Casal MN, Ota E. Nutrition-specific interventions for preventing and controlling anaemia throughout the life cycle: an overview of systematic reviews. Cochrane Database Syst Rev. 2021 Sep 26;9(9):CD013092. doi: 10.1002/14651858.CD013092.pub2. PMID 34564844